CLINICAL TRIAL: NCT05521386
Title: The Effects of Caffeine Supplementation on Heart Rate and Heart Rate Variability at Rest and During Submaximal Exercise
Brief Title: The Effects of Caffeine on Heart Rate and Heart Rate Variability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: StMarysUC5
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Caffeine
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine (Experimental): caffeine dose of 5 mg per kg of body mass administered orally via a gelatine capsule
  Interventions: Drug: Caffeine
- Placebo (Placebo Comparator): maltodextrin (placebo) dose of 5 mg per kg of body mass administered orally via a gelatine capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caffeine — Single pill in an acute dose of 5 mg per kg of body mass
  Arms: Caffeine
Drug: Placebo — Single pill in an acute dose of 5 mg per kg of body mass
  Arms: Placebo

SUMMARY:
In previous research we have shown that an acute caffeine dose of 5 mg/kg body mass reduces heart rate at rest and during low intensity exercise, with the effect dissipating as exercise intensity increases. If, as suspected, the effect at rest and at low intensities is due to an effect of caffeine on parasympathetic activity, this is likely to be reflected in an increase in heart rate variability (the beat-to-beat fluctuation in heart rate). The aim of this study is therefore to investigate the effect of caffeine on heart rate and heart rate variability at rest and during submaximal exercise.

ELIGIBILITY:
Inclusion Criteria:

* Trained cyclists

Exclusion Criteria:

* Injured or a contraindicative medical condition

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability | From baseline to completion, up to 31 days
  Change from baseline in heart rate variability measured at rest and at five different exercise intensities (40, 50, 60, 70 and 80% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer

SECONDARY OUTCOMES:
Heart rate | From baseline to completion, up to 31 days
  Change from baseline in heart rate measured at rest and at five different exercise intensities (40, 50, 60, 70 and 80% percent of maximal oxygen uptake) on an electromagnetically-braked cycle ergometer

REFERENCES:
- [Derived] Glaister M, Lythgoe D, Kamath S. The Effects of Caffeine on Heart Rate and Heart Rate Variability at Rest and During Submaximal Cycling Exercise. Res Q Exerc Sport. 2025 Mar;96(1):155-163. doi: 10.1080/02701367.2024.2377303. Epub 2024 Jul 15. PMID 39008947